CLINICAL TRIAL: NCT03584321
Title: A Multi-center, Retrospective, Registry Study to Estimate the Current Status of Patients With Non-Obstructive coroNary Artery Disease (CAD) Confirmed Via Coronary Angiography (CAG) (RESPOND Study)
Brief Title: Retrospective Study to Estimate the Current Status of Patients With Non-Obstructive coroNary Artery Disease
Acronym: RESPOND
Status: Completed | Type: Observational
Sponsor: Merck KGaA, Darmstadt, Germany (Industry)
Collaborators: Merck Serono Co., Ltd., China (Industry)
Responsible Party: Sponsor
Other Study IDs: MS200101_0003
Record Dates: First submitted 2018-06-29; First posted 2018-07-12 (Actual); Last update posted 2018-10-30 (Actual); Status verified 2018-10

CONDITIONS: Non-Obstructive Coronary Artery Disease
Keywords: Non-Obstructive Coronary Artery Disease; Coronary Angiography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Participants with Coronary Artery Disease: Participants with suspected or confirmed coronary artery disease who underwent coronary angiography during 01 Jan 2013 and 31 Dec 2015 will be observed in the study.

SUMMARY:
The study will estimate the current status of participants with non-obstructive coronary artery disease confirmed via coronary angiography.

ELIGIBILITY:
Inclusion Criteria:

* Participants who had typical or atypical angina symptom before Coronary Angiography examination
* Underwent CAG between 01 Jan 2013 and 31 Dec 2015
* Other protocol defined inclusion criteria could apply

Exclusion Criteria:

* Participant with history of percutaneous coronary intervention or coronary artery bypass surgery
* Participant with history of myocardial infarction
* Participant with history of cardiac transplant or valve surgery
* Presenting with Acute myocardial infarction for coronary angiography
* CAG showed myocardial bridge and coronary stenosis greater than or equal to 50 percent during systole period
* Incomplete or missing data in CAG report
* Other protocol defined exclusion criteria could apply

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Participants who were suspected or had confirmed coronary artery disease and who underwent coronary angiography between 01 Jan 2013 and 31 Dec 2015 will be observed in the study.
Sampling Method: Probability Sample
Enrollment: 1600 (Actual)
Dates: Start 2017-09-13 (Actual); Primary Completion 2018-07-11 (Actual); Study Completion 2018-07-11 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants with Non-Obstructive Coronary Artery Disease (CAD) | Up to 10 Months

SECONDARY OUTCOMES:
Percentage of Participants With Combined Cardiovascular Risk Factors | Up to 10 Months
  Combined cardiovascular risk factors include: body mass index, smoking habit, hypertension, hyperlipidemia diabetes mellitus, lack of exercise, alcohol intake and family history of early onset cardiovascular disease. Percentage of participants with combined cardiovascular risk factors will be reported.
Percentage of Participants With Angina Symptoms | Up to 10 months
Percentage of Participants With Pathologic Echocardiography Results | Up to 10 Months
Ventricular Wall thickness in Participants With Obstructive and Non-Obstructive Coronary Artery Disease (CAD) | Up to 10 Months
  Mean left ventricular posterior wall thickness (LVPW), interventricular septum (IVS) thickness, other ventricular wall thickness will be assessed for the participants with obstructive and non-obstructive CAD.
Left Ventricular End-Diastolic Volume (LVEDV) in Participants With Obstructive and Non-Obstructive Coronary Artery Disease (CAD) | Up to 10 Months
Left Ventricular End Diastolic Diameter (LVEDD) in Participants With Obstructive and Non-Obstructive Coronary Artery Disease (CAD) | Up to 10 Months
Ventricular Wall Motion in Participants With Obstructive and Non-Obstructive Coronary Artery Disease (CAD) | Up to 10 Months
Ratio of Early Trans-Mitral Flow (E) and Late Trans-Mitral Flow by Atrial Contraction (A) in Participants with Obstructive and Non-Obstructive Coronary Artery Disease (CAD) | Up to 10 Months
Left Ventricular Ejection Fraction (LVEF) in Participants with Obstructive and Non-Obstructive Coronary Artery Disease (CAD) | Up to 10 Months
Percentage of Participants Receiving Anti-ischemic Drugs | Up to 10 Months
Percentage of Participants with Myocardial Event Prevention | Up to 10 Months
  Percentage of participants achieving event prevention by antiplatelet agent, anticoagulants, β-blockers, Angiotensin converting enzyme inhibitor (ACEI), Angiotensin receptor blocker (ARB), statin, aldosterone antagonist will be reported.
Percentage of Participants With Obstructive and Non-Obstructive Coronary Artery Disease (CAD) Segregated by Age Groups, Genders, Races and Provinces | Up to 10 Months
Correlation Coefficient Between Participants With Non-obstructive CAD confirmed by CAG and Clinical Characteristics | Up to 10 Months
  Correlation coefficient between the participants with non-obstructive CAD and different clinical characteristics like demographic characteristics, combined cardiovascular risk factors and angina symptoms will be assessed using logistic regression analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — Merck Serono Co., Ltd, the biopharmaceutical division of Merck KGaA, Darmstadt, Germany
Locations (1):
- Please Contact the Merck KGaA Communication Center, Darmstadt, Germany

IPD SHARING:
Plan to Share IPD: No